CLINICAL TRIAL: NCT07132385
Title: Perimenopause: Window for Exercise and Resilience Pilot Study
Brief Title: Feasibility of Different Types of Exercise Training in Perimenopausal Females
Acronym: POWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSREB56686
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Women
Keywords: menopause; perimenopause; exercise
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: It is not possible to blind participants to their assigned intervention. Care providers are not involved. The outcome assessors for any assessments involving potential for subjectivity in data collection or analysis will be blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Guidelines-based moderate-intensity continuous exercise (Experimental): 150 weekly minutes of moderate-intensity aerobic activity
  Interventions: Behavioral: Guidelines-based moderate-intensity continuous exercise
- High-intensity interval training (Experimental): Periods of high intensity effort (1-4 min) interspersed with periods of rest (1-3 min)
  Interventions: Behavioral: High-intensity interval training
- Stretching exercise (Active Comparator): whole-body stretching
  Interventions: Behavioral: Stretching exercise

INTERVENTIONS:
Behavioral: Guidelines-based moderate-intensity continuous exercise — Through a combination of exercise trainer-led in-person and virtual sessions, participants will be guided to achieve 150 weekly minutes of moderate-intensity aerobic activity (total intervention is 6 weeks)
  Arms: Guidelines-based moderate-intensity continuous exercise
Behavioral: High-intensity interval training — Through a combination of exercise trainer-led in-person and virtual sessions, participants will be guided to achieve 75 weekly minutes of high-intensity interval training.
  Arms: High-intensity interval training
Behavioral: Stretching exercise — Twice weekly virtual instructor-led whole-body stretching class.
  Arms: Stretching exercise

SUMMARY:
Throughout the menopause transition, women experience many symptoms (i.e., hot flashes, night sweats) that can significantly reduce their quality of life. Moreover, their risk of heart disease increases substantially. The years before menopause called "perimenopause" present a critical window of intervention to alleviate menopause symptoms and improve health outcomes. Our team is therefore interested in comparing the potential benefits of different approaches including following the Health Canada guidelines (i.e., accumulating 150 min of moderate-to-vigorous aerobic physical activity weekly); performing high-intensity interval training (HIIT), which involves alternating periods of intense exercise with periods of rest; or stretching in perimenopause. As a first step towards this goal, this study will assess how easy and enjoyable the interventions are to follow over a 6-week period. The information gained from this study will be used to perform a larger study with enough participants to assess the health and quality of life impacts of adopting these different strategies in perimenopause.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of 3 groups and complete a 6 week intervention: 1) Moderate intensity continuous training (MICT) following the Health Canada guidelines (Group 1); 2) High-intensity interval training (HIIT) (Group 2); or 3) Stretching (Group 3). Before and after the intervention, participants will complete questionnaires to assess your menopause symptoms, stress levels and quality of life. Before and after the intervention the research team will also assess participants' body composition (fat mass and muscle mass) using a BodPod, and insulin sensitivity using an oral glucose tolerance testing with blood sampling. After the intervention, investigators will also ask that participants complete questionnaires that indicate how easy and enjoyable the intervention was to follow.

ELIGIBILITY:
Inclusion Criteria:

* Biological females in early and late perimenopause. Menopausal stage will be defined according to the Stages of Reproductive Aging Workshop +10 (STRAW+10). According to STRAW+10, perimenopause is characterized by menstrual cycle irregularity, specifically defined as having bleeding in the previous 12 months but at least a 7-day difference from usual menstrual cycle length
* Experiencing menopause symptoms (e.g., hot flashes, night sweats, joint stiffness)
* Aged 40 years or older
* Multiple risk factors for cardiometabolic disease, namely being sedentary (<30 min of moderate-vigorous physical activity/week), having a BMI ≥25 kg/m2, and a waist circumference indicative of abdominal obesity, specific to BMI (e.g., BMI 25-29.9: WC: 90cm; BMI 30-34.9: WC: 105cm; BMI 35-35.9: WC:115cm).

Exclusion Criteria:

* History of reproductive surgeries including oophorectomy, hysterectomy, ablation or gender-affirming.
* Diagnosis of cardiovascular disease, type 2 diabetes, non-alcoholic fatty liver disease, cancer (except for non-melanoma skin cancer), respiratory disease (e.g., Chronic Obstructive Pulmonary Disease or severe or uncontrolled asthma), uncontrolled hyper- or hypogonadism (change in medication or dosage in last 6 months and with major symptoms), and/or Polycystic Ovary Syndrome
* Major signs or symptoms (regardless of known diagnosis) of cardiovascular diseases, diabetes, or renal disease
* The use of medication that could impact blood glucose
* Pregnant or post-partum <12 months, lactating or breast feeding within 3 months of the start of study
* Recreational smoking (e.g., tobacco, smoking)
* Actively engaging in a low-carbohydrate diet (e.g., ketogenic, Atkins)
* Using transdermal hormones, taking exogenous hormones, or receiving exogenous hormones from other means (e.g., intrauterine device)
* Significant weight loss (i.e., >5 kg) in past 3 months or currently taking weight loss medications

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intervention Adherence | End of week 6
  Determined by the percentage of in-person and online sessions attended over those prescribed as well as exercise intensity adherence based on heart rate data collected via Garmin smartwatch
Enrolment | End of week 6
  Determined by the percentage of participants enrolled in study over those assessed for eligibility
Study Assessment Adherence | End of week 6
  Determined by the percentage of study assessments completed over those included as part of the study.
Attrition | End of week 6
  Determined by the percentage of participants who request withdrawal, are lost to follow-up, or experience injury preventing completion of the study over those enrolled
Intervention acceptability | End of week 6
  Assessed via an intervention-specific researcher-developed questionnaire

SECONDARY OUTCOMES:
Systemic insulin resistance | 6 weeks
  Systemic insulin resistance As assessed by the Matsuda Index calculated from an oral glucose tolerance test
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | Calculated as: (fasting insulin*fasting glucose)/22.5 6 weeks
  Calculated as: (fasting insulin*fasting glucose)/22.5
Cardiorespiratory fitness | 6 weeks
  Measured as peak volume of oxygen consumption via indirect calorimetry
Body circumferences | 6 weeks
  Waist and hip circumferences measured by inelastic tape
Whole-body fat and fat free mass | 6 weeks
  Measured by BodPod
Menopausal symptom presence and severity | 6 weeks
  Assessed by The Menopause-specific Quality of Life (MENQOL) questionnaire. The 29-item questionnaire measures four domains of symptoms (vasomotor, psychosocial, physical, sexual), capturing both their presence (yes/no) and severity (7-point Likert scale, where a higher score indicates a greater severity).
Sleep | 6 weeks
  Assessed by sleep time and efficiency via Garmin smartwatch as well as the Pittsburgh Sleep Quality Index (PSQI); score ranges from 0-21, with higher scores indicating poorer sleep quality
Depressive symptoms | 6 weeks
  Measured by the Patient Health Questionnaire-9 (PHQ-9), where individual scores range from 0-27, and the Beck Depression Inventory, where scores range from 0-63; for both measures, higher scores indicate greater depressive symptom severity
Health-related quality of life | 6 weeks
  Assessed by RAND-36, where an independent score is provided for 8 scales ranging from 0 to 100, with a higher score indicating better quality of life
Psychosocial stress | 6 weeks
  Assessed by the perceived stress scale where scores can range from 0 to 40, with higher scores indicating higher perceived stress
Anxiety symptoms | 6 weeks
  Measured by the Generalized Anxiety Disorder 7-item scale (GAD-7) where scores can range from 0-21, with higher scores indicating greater anxiety
Framingham 10-year risk (%) | 6 weeks
  Calculated using standardized scoring system
Systolic and Diastolic Blood pressure | 6 weeks
  Measured after several minutes of supine rest
Heart rate variability | 6 weeks
  Measured via electrocardiogram
Aortic stiffness (central) | 6 weeks
  Measured by pulse wave velocity using applanation tonometry
Brachial artery endothelial function | 6 weeks
  Measured via flow-mediated dilatation test
Dietary intake | 6 weeks
  Assessed via MyFitness Pal 3-day food records

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No